CLINICAL TRIAL: NCT01356810
Title: Manejo Ambiental Profilactico Del Delirium Intrahospitalario
Brief Title: Prophylactic Environmental Management of Delirium
Acronym: MAPDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Responsible Party: Principal Investigator, Felipe Martinez, Prophylactic Environmental Management of Delirium (MAPDI), Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P06/11
Record Dates: First submitted 2011-05-16; First posted 2011-05-20 (Estimated); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Delirium; Falls
Keywords: Delirium; Primary Prevention; Elderly
MeSH Terms: conditions — Delirium | interventions — Milieu Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard Care (Placebo Comparator): Delirium management defined by the attending physician.
  Interventions: Other: Standard Care
- Environmental Intervention (Experimental)
  Interventions: Other: Environmental Intervention

INTERVENTIONS:
Other: Environmental Intervention — The environmental intervention consisted of daily reorientation, avoidance of sensorial deprivation, longer visiting hours, the availability of a clock, a calendar and the presence of familiar objects in the room.
  Arms: Environmental Intervention
Other: Standard Care — Delirium management by the attending physician's preferences.
  Arms: Standard Care

SUMMARY:
Delirium is a complex neuropsychiatric syndrome with an acute onset and fluctuating course which is presented in 15 to 20% of patients admitted to general wards. It is a potentially life - threatening complication which can be prevented. It is the objective of this randomized controlled trial to evaluate whether a multicomponent environmental intervention could reduce the incidence of delirium in a general medical ward.

DETAILED DESCRIPTION:
A total of 287 patients 65 years of age or older who had been admitted to a general medicine ward and who were at risk of delirium were studied. Eligible patients were randomized to a multicomponent environmental intervention or standard care. Both groups were well balanced in patients characteristics and followed during the full hospital stay by a group trained in the application of the confusion assessment method to detect incident delirium.

ELIGIBILITY:
Inclusion Criteria:

* Above 65 years of age and one of the following:
* Age above 70 years.
* Alcoholism
* Cognitive deficit (Mini mental state examination <24 points)
* Metabolic disturbance (Hyponatremia, Hypernatremia, Hyperkalemia, Hypokalemia Hyperglycemia or Hypoglycemia)

Exclusion Criteria:

* Delirium at admission.
* Admittance to a ward other than general internal medicine.
* Lack of family support.
* Informed consent refusal.
* Hospitalization in a room with more than two beds.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 287 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Delirium | Daily during the entire hospital stay (Average: 10 days, Maximum: 42 days)
  New episodes of delirium during the hospital stay

SECONDARY OUTCOMES:
Incidence of Falls | Daily during the entire hospital stay (Average: 10 days, Maximum: 42 days
  New episodes of Falls

CONTACTS AND LOCATIONS:
Overall Officials: Felipe T Martinez, MD, Principal Investigator — Universidad de Valparaiso
Locations (1):
- Hospital Naval Almirante Nef, Viña del Mar, Región de Valparaíso, Chile